CLINICAL TRIAL: NCT02691052
Title: Non-interventional Study on Quality of Life, Efficacy and Tolerability of Nab-paclitaxel/Gemcitabine Firstline Therapy in Patients With Metastatic Pancreatic Cancer
Brief Title: Observational Study on Quality of Life of Patients Receiving Nab-paclitaxel/Gemcitabine First Line Therapy, Including a Translational Program
Acronym: QoliXane
Status: Completed | Type: Observational
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Trium Analysis Online GmbH (Industry); mca Berlin (Unknown)
Responsible Party: Sponsor
Other Study IDs: QoliXane
Record Dates: First submitted 2016-02-12; First posted 2016-02-25 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Tumor containing tissues are collected for a translational program focusing on defining prognostic and predictive factors.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pts receiving nab-paclitaxel/gemcitabine: Patients with metastatic pancreatic cancer undergoing a firstline therapy with nab-paclitaxel and gemcitabine will be asked to fill in an EORTC QLQ-C30 questionnaire and an additional questionnaire on worries about quality of life impairments every 4 weeks. No further intervention.
  Interventions: Other: Quality of Life questionnaire

INTERVENTIONS:
Other: Quality of Life questionnaire — EORTC QLQ-C30 questionnaire
  Other Names: EORTC QLQ-C30

SUMMARY:
Current studies resulted in a superiority of a combination of nab-paclitaxel and gemcitabine vs. gemcitabine mono therapy, but no data are available yet on the quality of life (QoL) under this combination therapy. In the framework of a German multicenter prospective, observational study ('QoliXane'), detailed QoL-data are now collected. QoL development under treatment will be analyzed and data will be compared to existing data of the gemcitabine mono therapy.

QoL and course of therapy are collected using the EORTC C30 questionnaires once a month over a 6-month period. Additionally patients are requested to answer a supplementary questionnaire addressing e.g. fears related to QoL deterioration and side effects of chemotherapy. Primary endpoint is the proportion of patients with maintained Global Health Status/QoL at 3 months (10 points threshold). 600 patients shall be enrolled at about 90 study sites in Germany.

ELIGIBILITY:
Inclusion Criteria:

* metastatic pancreatic carcinoma
* no previous therapy in the metastatic stage
* planned firstline therapy with nab-paclitaxel and gemcitabine

Exclusion Criteria:

* previous therapy in the metastatic stage
* patient unable to understand the study and to give informed consent
* patient unable to answer quality of life questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic pancreatic cancer subject to firstline therapy with nab-paclitaxel and gemcitabine
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-12; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Global Health Status/Quality of Life Score at 3 months | 3 months
  Rate of patients without deterioration of their global health status/quality of life score according to EORTC QLQ-C30 after 3 months

SECONDARY OUTCOMES:
Global Health Status/Quality of Life Score at 6 months | 6 months
  Rate of patients with an improvement of their global health status/quality of life score according to EORTC QLQ-C30 after 6 months
Limited Baseline Condition | 3 and 6 months
  Rate of patients with a limited baseline general condition (ECOG 2 or 3) and stable or improved Global Health Status/Quality of Life Score after 3 and 6 months
Therapy effects on Global Health Status/Quality of Life Score | 3 months
  Effect of therapy on Global Health Status/Quality of Life Score and other symptoms and scales assessed by EORTC QLQ-C30: rate of patients with improved, stable or deteriorated score
Prognostic validity of Global Health Status/Quality of Life Score as assessed by tumor response and EORTC QLQ-C30 | 6 months
Median time until definitive deterioration of Global Health Status/Quality of Life Score and other functional and symptom scales of EORTC QLQ-C30 | 6 months
Influence of Neuropathy on Quality of Life compared to other treatment-related adverse events as assessed by CTCAE v4.0 | 6 months
Comparison of Global Health/Quality of Life scores as assessed by EORTC QLQ-C30 to historical Global Health/Quality of Life score data of gemcitabine mono-therapy | 6 months
Tumor response (RECIST) | 6 months
Progression free survival as assessed by tumor response | 6 months
Overall survival as assessed by survival data one year after patient enrollment | 1 year
Efficacy in high ECOG and high bilirubin patients | 6 months
Adverse events | 6 months
Adverse events in special subgroups like high ECOG or high bilirubin patients | 6 months
Correlations of tumor response and survival with genetic alterations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Institute of Clinical Cancer Research
Locations (1):
- Krankenhaus Nordwest gGmbH - Institute of Clinical Cancer Research, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Al-Batran SE, Hofheinz RD, Reichart A, Pauligk C, Schonherr C, Schlag R, Siegler G, Dorfel S, Koenigsmann M, Zahn MO, Schubert J, Aldaoud A, Hoffkes HG, Schulz H, Hahn L, Uhlig J, Blau W, Stauch M, Weniger J, Wolf M, Jacobasch L, Bildat S, Wehmeyer J, Homann N, Trojan J, Waidmann O, Fietz T, Feustel HP, Groschek M, Wierecky J, Waibel K, Mahlmann S, Schwindel U, Peters U, Schuch G, Pink D, Eschenburg H, Worns MA, Harich HD, von Weikersthal LF, Dassler KU, Behringer DM, Messmann H, Kretzschmar A, Gallmeier E, Forstbauer H, Kunzmann V, Papke J, Buchner-Steudel P, Vehling-Kaiser U, Springfeld C, Vogel A, Ettrich TJ, Schaaf M, Hausen GZ, Gotze TO; Arbeitsgemeinschaft Internistische Onkologie (AIO). Quality of life and outcome of patients with metastatic pancreatic cancer receiving first-line chemotherapy with nab-paclitaxel and gemcitabine: Real-life results from the prospective QOLIXANE trial of the Platform for Outcome, Quality of Life and Translational Research on Pancreatic Cancer registry. Int J Cancer. 2021 Mar 15;148(6):1478-1488. doi: 10.1002/ijc.33336. Epub 2020 Oct 23. PMID 33038277